CLINICAL TRIAL: NCT06437678
Title: A Single-Center, Prospective Phase II Clinical Study of Liposomal Irinotecan Monotherapy for Third-Line and Beyond Recurrent/Refractory Advanced Gastric Cancer
Brief Title: Phase II Study of Liposomal Irinotecan for Advanced Refractory Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-498
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent/Refractory Advanced Gastric Cancer (Other)
  Interventions: Drug: Liposomal Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Liposomal Irinotecan Hydrochloride — Liposomal Irinotecan Hydrochloride Injection (Ⅱ) 56.5mg/m2 every 2 weeks

SUMMARY:
To evaluate the objective response rate (ORR) and disease control rate (DCR) of liposomal irinotecan monotherapy in the treatment of recurrent/refractory advanced gastric cancer.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, prospective clinical trial aimed at evaluating the efficacy and safety of liposomal irinotecan monotherapy in the treatment of recurrent/refractory advanced gastric cancer. The study targets patients with locally advanced, recurrent, or metastatic/previous treatment-refractory adenocarcinoma of the stomach or gastroesophageal junction. The primary endpoints of the study are objective response rate (ORR) and disease control rate (DCR). It plans to enroll 50 patients with locally advanced, recurrent, or metastatic/previous treatment-refractory adenocarcinoma of the stomach or gastroesophageal junction. Subjects will sign informed consent and undergo screening for eligibility before enrollment. Subjects will receive the following treatment: Liposomal Irinotecan Hydrochloride Injection (Ⅱ) 56.5mg/m2 every 2 weeks. Safety visits will be conducted on Day 1 of each treatment cycle, at the end of the study treatment, and 30 days (±7 days) after the end of the study treatment. Imaging assessments will be performed according to RECIST 1.1 criteria, including chest CT, enhanced CT scans of the abdomen and pelvis, or chest CT plain scan plus abdominal/pelvic MRI scan for patients allergic to contrast agents. Suspected cases of brain metastases will require brain enhanced MRI or enhanced CT. Bone scan examination will be conducted if bone metastases are suspected clinically or radiologically. Patients who discontinue treatment due to reasons other than radiological progression during the treatment period will undergo imaging examination at the end of treatment unless it has been conducted within 28 days. Subjects will undergo survival follow-up every 3 months after the end of treatment to collect and record survival status and subsequent anti-tumor treatment until death or loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join this study and sign an informed consent form;
* Age ≥18 years and ≤75 years;
* Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma;
* CT or biopsy-confirmed recurrent or metastatic gastric or gastroesophageal junction adenocarcinoma;
* Previously received at least one line of standard first- and second-line therapy (e.g., chemotherapy, targeted therapy), and experienced disease progression or intolerance;
* Interval of ≥4 weeks since previous chemotherapy, immunotherapy, or radiotherapy;
* Expected survival of ≥12 weeks;
* ECOG performance status score of 0-2;
* Normal major organ function, meeting the following criteria:

  1. Hematologic criteria:

     (No blood transfusion or blood products, and no use of G-CSF or other hematopoietic growth factors within 14 days) Absolute neutrophil count ≥1.5×10^9/L; Platelets ≥80×10^9/L; Hemoglobin ≥80 g/L.
  2. Biochemical criteria:

     Total bilirubin <1.5×ULN; ALT and AST ≤2.5×ULN (without liver metastasis) / ALT and AST ≤5×ULN (with liver metastasis); Serum creatinine ≤1.5×ULN or creatinine clearance >50 ml/min (Male: creatinine clearance = ((140 - age) × weight) / (72 × serum creatinine); Female: creatinine clearance = ((140 - age) × weight) / (72 × serum creatinine) × 0.85; weight in kg; serum creatinine in mg/mL).
  3. Urine protein (semi-quantitative method) less than 2+;
  4. Normal coagulation function (including INR, APTT, PT, FIB).
* Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and agree to use effective contraception during the study and for 120 days after the last dose. Male participants with partners of childbearing potential must be surgically sterilized or agree to use effective contraception during the study and for 120 days after the last dose.

Exclusion Criteria:

* Having a history of or currently suffering from other malignant tumors;
* Previous or current use of irinotecan drugs;
* Having any chronic or significant disease deemed intolerable to treatment (e.g., severe heart disease, uncontrolled hypertension, significant liver or kidney dysfunction, etc.);
* History of gastrointestinal perforation, abdominal abscess, or recent (within 3 months) bowel obstruction, or imaging or clinical symptoms indicating the presence of bowel obstruction;
* Significant clinically relevant bleeding symptoms or a clear tendency to bleed within 3 months before the first dose of the study drug, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis; if fecal occult blood is positive at baseline, retesting is allowed. If retesting remains positive, a gastroscopy is required (unless gastroscopy has been performed within the past 3 months to exclude these conditions);
* Currently undergoing treatment for an active infection (e.g., requiring antibacterial, antiviral, or antifungal therapy);
* Active hepatitis (Hepatitis B: HBsAg positive and HBV DNA ≥500 IU/ml; Hepatitis C: HCV antibody positive and HCV RNA > upper limit of normal);
* Congenital or acquired immunodeficiency (e.g., HIV infection);
* Suffering from a mental illness that could interfere with consent or follow-up;
* Having any active autoimmune disease or a history of autoimmune disease with a risk of recurrence;
* Planned or previous organ or allogeneic bone marrow transplantation;
* Currently having interstitial pneumonia or interstitial lung disease, a history of interstitial pneumonia or interstitial lung disease requiring steroid treatment, or a screening CT showing active pneumonia or severe lung dysfunction; active tuberculosis;
* Currently using or recently used immunosuppressive drugs or systemic corticosteroids for immunosuppressive purposes;
* Received an attenuated live vaccine within 28 days before the first dose of the study drug, or requires such a vaccine during the treatment period or within 60 days after the last dose;
* Known allergy to any study drug or excipients;
* Breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 1 year
  After treatment, the proportion of cancer patients whose tumors have shrunk to a predetermined value and can maintain the minimum time limit requirement is the sum of the complete response (CR) and partial response (PR) ratios.
Disease Control Rate (DCR) | through study completion, an average of 1 year
  The percentage of evaluable cases in cancer patients who have improved their condition (CR+PR) and stabilized their condition (SD) after treatment.

SECONDARY OUTCOMES:
OS (Overall survival) | Assessed up to 60 months
  The time between the date of enrollment and death caused by any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No